CLINICAL TRIAL: NCT00578409
Title: Identification of Predictive Factors for Survival of Patients With Recurrent Prostate Cancer From Clinical Features, Tissue Image Features and Molecular Biomarker Data
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Aureon Biosciences, Inc. (Industry); NYU MEDICAL CENTER (Unknown)
Responsible Party: Sponsor
Other Study IDs: 04-062
Record Dates: First submitted 2007-12-19; First posted 2007-12-21 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: Prostate Cancer
Keywords: castration resistant prostate cancer; progressive castrate metastatic prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — In a first analytical step, using only the clinical and pathological variables used in the original clinical mets castrate disease nomogram as inputs, supervised multivariate analytical techniques (SMA) were used to generate a new predictive model for patient survival. A similar approach will then be used to analyze a second group of approximately 223 pts in the state of a rising PSA14 after surgery or radiation therapy treated on a sequential series of IRB approved trials testing conjugate vaccines also consented on IRB protocol 90-40.

SUMMARY:
We seek to improve the predictive accuracy of the nomogram to predict survival for patients with castrate mets disease through the addition of pathological data, the results of automated machine vision based image analysis of H&E stained tumor tissue developed at Aureon Biosciences,and molecular biomarker studies (25 markers) determined by immunohistochemistry on tissue microarrays prepared from paraffin-embedded tumor.

ELIGIBILITY:
Inclusion Criteria:

Patients in the first retrospective study (Stage 1) must be part of the 409 patient strong MSKCC cohort with progressive metastatic prostate cancer which was used for the generation of the original nomogram.

For details please see original publication by Smaletz et al. Patients involved in the second retrospective study (Stage 2) must be part of the 223 patients with a rising PSA after surgery or radiation therapy who were treated on conjugate vaccine trials at MSKCC..

Exclusion Criteria:

For details of excluded patients on the clinical metastases castrate disease study, please see original publication by Smaletz et al.4

• (MSKCC - add reference if publication available for rising PSA patients)

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Stage 1 - Population: Progressive Metastatic Disease Stage 2 - Population: Rising PSA
Sampling Method: Non-Probability Sample
Enrollment: 758 (Actual)
Dates: Start 2004-05; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
The analysis for the progressive castrate mets disease population consists of two analytical steps. The first step involved the development of a predictive model of pt survival using supervised multivariate analytical (SMA)techniques | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Howard I Scher, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Web Site — http://www.mskcc.org